CLINICAL TRIAL: NCT04231669
Title: Intervention to Improve Developmental and Health Outcomes for Female Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Ghana (Other); BasicNeeds Ghana (Other); BIBIR Ghana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21HD099508 (NIH)
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Independent Child Migration
Keywords: child migration; child labor; sub-Saharan Africa; female adolescents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: bolstered care (No Intervention): Female adolescents in the bolstered care will receive services/education as usual in their respective schools. The usual care will be bolstered by providing school notebooks and lunch in the control arm (bolstered care will also be provided to treatment arm). Primary school education is universal and free in Ghana. Yet notebooks and lunch are costly expenses for families that create a barrier to school attendance. Hence, these will be provided to participants in all study schools.
- Anzansi Family Program (Experimental): In addition to bolstered care, participants(adolescent girls and caregivers) in this arm will receive the ANZANSI that combines Family Economic Empowerment (EE) with Multiple Family Groups (MFG).
  Interventions: Behavioral: Anzansi Family Program

INTERVENTIONS:
Behavioral: Anzansi Family Program — the ANZANSI that combines Family Economic Empowerment (EE) with Multiple Family Groups (MFG). Family EE includes: 1) Workshops on asset building, future planning, and protection from risks; 2) Child Development Account (CDA); and 3) Family income-generating/microenterprise promotion (IGA) component:
  MFG a family-centered, group-delivered, evidence-informed intervention designed for children and adolescents whose families struggle with poverty and associated stressors. The MFG is based on building family support through opportunities for parents and children to communicate in a safe setting with other families who have shared experiences, and allow each family to learn from one another. MFG builds protective factors for healthy parent-child relationships while addressing familial, social and community stressors and barriers to adolescent girls' well-being. Both adolecsnt girls and their caregivers will receive the intervention.
  Arms: Anzansi Family Program

SUMMARY:
The primary goal of this pilot study (R21) is to address the urgent need for theoretically and empirically informed interventions that prevent poor female youth's rural-to-urban migration for child labor in low and middle-income countries. The study will address the following specific aims: Aim 1: Pilot test the (i) feasibility and acceptability of ANZANSI; and (ii) preliminary impact of ANZANSI by comparing the control arm to the treatment arm on specific child development outcomes; Aim 2: Explore multi- level factors (individual, family, and programmatic) impacting participation in and experiences with the ANZANSI.

DETAILED DESCRIPTION:
The primary goal of this pilot study (R21) is to address the urgent need for theoretically and empirically informed interventions that prevent poor female youth's rural-to-urban migration for child labor in low and middle-income countries. The International Labor Organization (ILO) estimates that 11% of children (ages 5 to 17) worldwide are child laborers. ILO recently drew attention to migrant child laborers as an underreported, but more vulnerable group to adverse outcomes relative to children working locally. Sub-Saharan Africa (SSA) continues to be the continent with the highest rates of child labor, with Ghana registering one of the highest incidence rates at 22%, including unaccompanied child migrants engaged in labor. Adolescent girls make up the majority of unaccompanied rural-to-urban migrants in search of better economic opportunities. Studies document the myriad of serious threats to health and emotional well-being experienced by female adolescent migrants engaged in child labor. These threats underline the urgent need for theoretically-informed preventive interventions, specifically tailored to address the root causes of female child migrant labor and the needs of girls from economically insecure families and communities. Hence, this application titled ANZANSI Family Program focuses on girls before they drop out of school, but as they begin exhibiting possibility of dropping out. Specifically, ANZANSI is an innovative combination intervention program, combining an evidence-informed family-level economic empowerment (EE) aimed at creating and strengthening financial stability through the use of matched children savings accounts (CSA) and microfinance in poor households with a multiple family group (MFG) intervention addressing family functioning and parental beliefs around gender and child labor/ education. Informed by asset theory, parental ethnotheories framework; and the investigative team's research in SSA on child-wellbeing and poverty, the study uses a cluster randomized control design (N=10 schools; n=100 girls ages 11-14 at risk of dropping out of school and their caregivers), assigned to two study conditions (N= 5 schools; n=50 children at risk of dropping out of school and their caregivers in each condition). The control group will receive bolstered usual care, including books and school lunch and treatment group will receive a combination intervention (Family EE+MFG) called ANZANSI, to address the following specific aims: Aim 1: Pilot test the (i) feasibility and acceptability of ANZANSI; and (ii) preliminary impact of ANZANSI by comparing the control arm to the treatment arm on specific child development outcomes; Aim 2: Explore multi- level factors (individual, family, and programmatic) impacting participation in and experiences with the ANZANSI. This study is aligned with NICHD's mission to support research relevant to the psychological, behavioral, and educational development and health of children worldwide. Ultimately, our findings may guide approaches to address youth's unaccompanied rural-to-urban migration and involvement in child labor in SSA, and the associated negative consequences.

ELIGIBILITY:
Inclusion Criteria:

Adolescent girls' inclusion criteria are:

* Enrolled in school and living within a family (defined broadly -not necessarily biological parents)
* Ages 11 to 14
* Capable of giving assent
* Skipping school in the past academic term (with at least 10% of unexcused absences).

The caregiver inclusion criteria are:

* Self-identified as primary caregiver of the adolescent girl
* Capable of providing informed consent.

Exclusion Criteria:

* Participants (girls and caregivers) that do not meet the criteria or exhibit a lack of understanding of the study procedures and hence not able to provide informed consent will be excluded.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ghana, Accra, Ghana

REFERENCES:
- [Derived] Sensoy Bahar O, Ssewamala FM, Ibrahim A, Boateng A, Nabunya P, Neilands TB, Asampong E, McKay MM. Anzansi family program: a study protocol for a combination intervention addressing developmental and health outcomes for adolescent girls at risk of unaccompanied migration. Pilot Feasibility Stud. 2020 Dec 7;6(1):190. doi: 10.1186/s40814-020-00737-4. PMID 33372647

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: schools
Groups:
- Anzansi Family Program: In addition to bolstered care, participants in this arm will receive the ANZANSI that combines Family Economic Empowerment (EE) with Multiple Family Groups (MFG).
  Anzansi Family Program: the ANZANSI that combines Family Economic Empowerment (EE) with Multiple Family Groups (MFG). Family EE includes: 1) Workshops on asset building, future planning, and protection from risks; 2) Child Development Account (CDA); and 3) Family income-generating/microenterprise promotion (IGA) component:
  MFG a family-centered, group-delivered, evidence-informed intervention designed for children and adolescents whose families struggle with poverty and associated stressors. The MFG is based on building family support through opportunities for parents and children to communicate in a safe setting with other families who have shared experiences, and allow each family to learn from one another. MFG builds protective factors for healthy parent-child relationships while addressing familial, social and community stressors and barriers to adolescent girls' well-being.
Period: Overall Study
Arm/Group | Control: Bolstered Care | Anzansi Family Program
Started | 100; 5 schools | 100; 5 schools
Completed | 100; 5 schools | 94; 5 schools
Not Completed | 0; 0 schools | 6; 0 schools

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control: Bolstered Care | Anzansi Family Program | Total
Number analyzed (Participants) | 100 | 94 | 194
Age, Categorical [Count of Participants; unit: Participants] — Population: The numbers reported in the overall number of baseline participants correspond to caregivers and adolescents together.
  Participants
    adolescents: number analyzed (Participants) | 50 | 47 | 97
    adolescents: <=18 years | 50 | 47 | 97
    adolescents: Between 18 and 65 years | 0 | 0 | 0
    adolescents: >=65 years | 0 | 0 | 0
    caregivers: number analyzed (Participants) | 50 | 47 | 97
    caregivers: <=18 years | 0 | 0 | 0
    caregivers: Between 18 and 65 years | 48 | 46 | 94
    caregivers: >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The total number is the sum of caregivers and adolescent girls.
  Participants
    adolescents: number analyzed (Participants) | 50 | 47 | 97
    adolescents: Female | 50 | 47 | 97
    adolescents: Male | 0 | 0 | 0
    caregivers: number analyzed (Participants) | 50 | 47 | 97
    caregivers: Female | 27 | 30 | 57
    caregivers: Male | 23 | 17 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Intention to Migrate
Description: Change in intention to migrate will be measured by one question: How likely do you (the adolescent girl) see yourself migrating? The question uses a likert scale ranging from 1 (very unlikely) to 5 (very likely).
Time Frame: Baseline, post-test (9 months), 6-months follow-up
Population: Adolescent girls. One participant was lost to follow-up at 9 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control: Bolstered Care | Anzansi Family Program
Number analyzed (Participants) | 50 | 47
Score on a scale
  6-months follow-up | 1.72 (1.21) | 1.15 (0.751)
  post-test (9 months): number analyzed (Participants) | 50 | 46
  post-test (9 months) | 1.42 (0.84) | 1.28 (0.72)
  Baseline | 1.6 (1.05) | 1.64 (1.21)
Statistical Analysis 1: Comparison: Control: Bolstered Care vs Anzansi Family Program; Test type: Superiority; p = 0.05, Linear Mixed-effects regression

2. Secondary Outcome: Attitudes Towards School
Description: Change in attitudes towards school were measured by School attitude assessment survey (SAAS; McCoach, 2002). The survey consists of 20 items rated on a 5-point Likert scale (1 = not at all, 2 = a little bit, 3 = pretty well, 4 = well, and 5 = very well; range 20 to 100). The scale measures aspects of students' lives that predict their academic achievement, including peer attitudes, attitudes toward school, self-motivation, and self-regulation. The items were coded and summed, with the higher values representing higher positive attitudes toward school (Cronbach's alpha = 0.92).
Time Frame: baseline, post-test (9 month), 6 month follow-up (6-month post intervention completion)
Population: Adolescent girls. One participant was lost to follow-up at 9 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treatment Arm: Treatment arm (ANZANSI family program). The ANZANSI family program combined two evidence-based interventions previously tested in the SSA: the Family Economic Empowerment (FEE) intervention to enhance household financial stability and the Multiple Family Group (MFG) to strengthen family relations and address cultural norms.
- Control Arm: Control arm (Bolstered usual care). Adolescent girls in the control arm received educational services from their schools, supplemented with additional resources, including school textbooks and lunch (the same resources were provided to the treatment group). Although primary education in Ghana is universally accessible and free, the costs associated with essential items such as notebooks and meals pose significant challenges for families and can hinder regular school attendance. To address this, study participants across all schools received these supplementary materials to support their education.
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 50
score on a scale
  6 month follow-up | 90.23 (6.83) | 85.12 (9.64)
  post-test (9 month: number analyzed (Participants) | 46 | 50
  post-test (9 month | 80.28 (10.46) | 75.9 (10.85)
  Baseline | 87.47 (10.61) | 84.76 (9.46)

3. Secondary Outcome: School Attendance
Description: Change in school attendance will be measured by school attendance reports. Number of missed days will be collected
Time Frame: baseline, post-test (9 month), 6 month follow-up (6-month post intervention completion)
Population: This outcome only applies to adolescent girls.
Measure: Count of Participants; unit: Participants
Groups:
- Anzansi Family Program: In addition to bolstered care, participants(adolescent girls and caregivers) in this arm will receive the ANZANSI that combines Family Economic Empowerment (EE) with Multiple Family Groups (MFG).
  Anzansi Family Program: the ANZANSI that combines Family Economic Empowerment (EE) with Multiple Family Groups (MFG). Family EE includes: 1) Workshops on asset building, future planning, and protection from risks; 2) Child Development Account (CDA); and 3) Family income-generating/microenterprise promotion (IGA) component:
  MFG a family-centered, group-delivered, evidence-informed intervention designed for children and adolescents whose families struggle with poverty and associated stressors. The MFG is based on building family support through opportunities for parents and children to communicate in a safe setting with other families who have shared experiences, and allow each family to learn from one another. MFG builds protective factors for healthy parent-child relationships while addressing familial, social and community stressors and barriers to adolescent girls' well-being. Both adolecsnt girls and their caregivers will receive the intervention.
Arm/Group | Control: Bolstered Care | Anzansi Family Program
Number analyzed (Participants) | 50 | 47
Participants
  Baseline Baseline: Less than 10% | 23 | 20
  Baseline Baseline: Equal to or more than 10% | 27 | 27
  post-test: Less than 10% | 24 | 27
  post-test: Equal to or more than 10% | 26 | 20
  6-month follow-up: Less than 10% | 27 | 32
  6-month follow-up: Equal to or more than 10% | 23 | 15

4. Secondary Outcome: Self-concept
Description: Change in self-concept was measured by the Tennessee Self-Concept Scale Short Form (TSCS). The 20-item short version of the original 100-item TSCS scale assesses adolescents' perception of self-identity and self-satisfaction. The items are rated on a 5-point Likert scale ranging from 1 = always false to 5 = always true. The theoretical range for the TSCS is 20-100, with higher scores representing a more positive self-concept.
Time Frame: baseline, post-test (9 months), 6 month follow-up (6-month post intervention completion)
Population: Adolescent girls. One participant was lost to follow-up at 9 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 50
score on a scale
  6-months follow-up | 73.09 (9.17) | 72.74 (9.78)
  post-test (9 months): number analyzed (Participants) | 46 | 50
  post-test (9 months) | 76.5 (10.92) | 74.94 (12.58)
  Baseline | 80.36 (9.94) | 81.02 (7.83)

5. Secondary Outcome: Multidimensional Student Life Satisfaction
Description: change in life satisfaction was measured by Multidimensional Student Life Satisfaction Scale (MSLSS) (Wilson, 2015). The scale includes 40 items assessing life satisfaction on 5 specific aspects while maintaining an overall life satisfaction score (Huebner et al., 1998). Responses are rated on a 6-point Likert scale with 1 = strongly disagree, 2 = moderately disagree, 3 = slightly disagree, 4 = slightly agree, 5 = moderately agree, and 6 = strongly agree (theoretical range 40-240). To avoid the potential for type I error, the total score was summed up and used in the analysis, with the higher values representing higher satisfaction in student life.
Time Frame: baseline, post-test (9 months), 6 month follow-up (6-month post intervention completion)
Population: Adolescent girls. One participant was lost to follow-up at 9 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 50
score on a scale
  6 month follow-up | 189.83 (19.48) | 183.24 (21.15)
  post-test (9 months): number analyzed (Participants) | 46 | 50
  post-test (9 months) | 191.74 (23.42) | 182.92 (23.82)
  Baseline | 189.49 (15.20) | 186.98 (15.75)

6. Secondary Outcome: The Adolescent Stress Questionnaire (ASQ)
Description: Change in stress levels was measured by the Adolescent Stress Questionnaire (ASQ) (Byrne et al., 2007). The ASQ consists of 48 items, each measuring different stressors on a 5-point Likert scale ranging from 1 (not at all stressful) to 5 (very stressful). The questionnaire includes eight subscales: stress of home, stress of school performance, stress of school attendance, stress of peer pressure, stress of teacher interaction, stress about future uncertainty, stress of school or leisure conflict, and stress of financial pressure. We calculated a composite score by summing the responses, with higher scores indicating greater stress levels (theoretical range 48-240).
Time Frame: baseline, post-test (9 months), 6 month follow-up (6-month post intervention completion)
Population: Adolescent girls. One participant was lost to follow-up at 9 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 50
score on a scale
  6 month follow-up | 174.34 (38.37) | 163.84 (42.70)
  post-test (9 months): number analyzed (Participants) | 46 | 50
  post-test (9 months) | 148.52 (49.30) | 164.48 (37.56)
  Baseline | 113.40 (46.97) | 117.38 (56.15)

7. Secondary Outcome: Family Cohesion
Description: We assessed family cohesion using seven items (theoretical range: 7-35, Cronbach alpha = 0.84) adapted from both the Family Environment Scale (Moos, 1994) and the Family Assessment Measure (Skinner et al., 1983). The items measured the degree of commitment, help and support family members provide for one another. Participants were asked to rate how often each item occurred in their family using a 5-point scale (with 1 = 'never' and 5 = 'always'). Items included 'Do your family members ask each other for help before asking nonfamily members for help?', and 'Do you listen to what other family members have to say, even when you disagree?' Summary scores were created, with higher scores indicating higher levels of family cohesion.
Time Frame: baseline, post-test (9 months), 6 month follow-up (6-month post intervention completion)
Population: Adolescent girls. One participant was lost to follow-up at 9 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 50
score on a scale
  Baseline | 26.55 (6.74) | 28.34 (6.40)
  post-test (9 months): number analyzed (Participants) | 46 | 50
  post-test (9 months) | 30.98 (5.52) | 27.5 (6.36)
  6 month follow-up | 29.57 (7.12) | 29.04 (6.04)

8. Secondary Outcome: Child-caregiver Relationship
Description: The perceived child-caregiver relationship scale was adapted from the Family Assessment measure and assessed relationships on two dimensions: (1) acceptance and warmth - the extent to which the caregiver perceives as involved in their child's life; and (2) psychological autonomy - the extent to which the caregiver employs a non-coercive, democratic discipline and encourages the child to express individuality within the family. Participants were asked to rate the adults they live with, on each of the 16 items (range: 16-80), on a 5-point scale (1 = 'never' and 5 = 'always'). Sample items include: "Can you count on your parents to help her if she has a problem?" and "Do your parents keep challenging you to do the best in whatever you do?" Summary mean scores were created, with higher scores indicating a more positive child-caregiver relationship.
Time Frame: baseline, post-test (9 months), 6 month follow-up (6-month post intervention completion)
Population: We analyzed adolescent participant data. One participant was lost to follow-up at 9 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Bolstered Care | Anzansi Family Program
Number analyzed (Participants) | 50 | 47
score on a scale
  Baseline data | 61.92 (8.82) | 61.40 (10.01)
  post-test (9 months): number analyzed (Participants) | 50 | 46
  post-test (9 months) | 60.44 (6.14) | 62.98 (6.74)
  6 month follow-up (6-month post intervention completion) | 60.56 (6.38) | 61.45 (4.27)

9. Secondary Outcome: Social Support
Description: Change in social support was measured by the Social Support Behavior Scale. The SS-B measure consists of 45 items designed to tap five modes of support: emotional support, socializing, practical assistance, financial assistance, and advice/guidance. The Likert scale is from 1=strongly disagree to 5=strongly agree. The theoretical range is 45-225, with higher scores indicating higher social support.
Time Frame: baseline, post-test (9 months), 6 month follow-up (6-month post intervention completion)
Population: Adolescent data were analyzed from baseline to 15 months. One participant was lost to follow-up at 9 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Bolstered Care | Anzansi Family Program
Number analyzed (Participants) | 50 | 47
score on a scale
  Baseline | 163.26 (26.53) | 149.83 (30.0)
  post-test (9 months): number analyzed (Participants) | 50 | 46
  post-test (9 months) | 171.43 (21.99) | 183.5 (17.74)
  6 month follow-up (6-month post intervention completion) | 164.44 (23.30) | 183.28 (22.95)

10. Secondary Outcome: Perceived Social Support
Description: Change in perceived social support was measured by the Multidimensional Scale of Perceived Social Support. The MSPSS is a self-report measure to assess participants' social support. The 12-item scale had statements such as, "there is a special person who is around when I am in need," rated on a 5-point Likert scale ranging from strongly agree to strongly disagree, with 5=strongly agree, 4=agree, 3=neutral, 2=disagree, 1=strongly disagree.
  Responses were coded and added up. The theoretical range was 12-60, with higher scores indicating greater social support.
Time Frame: baseline, post-test (9 months), 6 month follow-up (6-month post intervention completion)
Population: Adolescent girls. One participant was lost to follow-up at 9 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 50
score on a scale
  6 month follow-up | 36.62 (3.75) | 34.32 (5.68)
  post-test (9 months),: number analyzed (Participants) | 46 | 50
  post-test (9 months), | 35.54 (4.11) | 30.18 (6.38)
  Baseline | 32.51 (4.86) | 32.32 (4.44)

11. Secondary Outcome: Gender Attitudes
Description: We assessed gender norms among caregivers using a 10-item scale adapted from the Gender Norm Attitudes Scale (Waszak et al., 2001), which measures participants' understanding of the appropriateness of behaviors as they relate to being female and male. The items in the scale encompass aspects related to educational performance, future expectations for both genders, family support, encouragement, decision-making, and involvement in intimate relationships and behaviors. The scale items featured binary responses (Agree = 1 and Disagree = 0). To create a summation score, items in the reverse direction were appropriately reverse-coded (theoretical range 0-10). Higher scores denote more egalitarian gender norms and beliefs.
Time Frame: baseline, post-test (9 months), 6 month follow-up (6-month post intervention completion)
Population: Caregiver data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Bolstered Care | Anzansi Family Program
Number analyzed (Participants) | 50 | 47
score on a scale
  6 month follow-up | 2.7 (2.18) | 3.04 (1.77)
  post-test (9 months): number analyzed (Participants) | 50 | 46
  post-test (9 months) | 2.84 (2.72) | 3.39 (2.91)
  Baseline | 2.06 (2.19) | 2.44 (2.17)

12. Secondary Outcome: Savings
Description: the average bank savings as measured by Bank statements
Time Frame: post-test (9 months)
Population: We analyzed bank savings information from the ANZANSI group. The control group had no bank data. We report the average bank savings for only the ANZANSI Family Program at 9 months in Ghana Cedis.
Measure: Mean (Standard Deviation); unit: Ghana cedis
Arm/Group | Control: Bolstered Care | Anzansi Family Program
Number analyzed (Participants) | 0 | 47
Ghana cedis |  | 401 (175)

13. Secondary Outcome: Future Orientation
Description: Change in future orientation was measured by two items evaluating adolescents' expectations and optimism regarding their educational goals. The first item asked participants, How sure are you that you will achieve your educational plans? with response options ranging from 1 = Not at all sure to 5 = Extremely sure. The second item asked, How hopeful are you that you will achieve your educational plans? with parallel response options ranging from 1 = Not at all hopeful to 5 = Extremely hopeful (theoretical range 2-10). For both items, higher scores indicated greater perceived likelihood of achieving educational goals and stronger optimism about the future. A composite future orientation score was created by summing the two items, with higher scores reflecting greater optimism and confidence in achieving educational aspirations. Only participants with non-missing values for both items were included in the composite measure.
Time Frame: baseline, post-test (9 months), 6 month follow-up (6-month post intervention completion)
Population: Adolescent Change in future orientation will be measured by the Thinking about the future measure. One participant was lost to follow-up at 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Bolstered Care | Anzansi Family Program
Number analyzed (Participants) | 50 | 47
score on a scale
  Baseline | 8.34 (1.49) | 8.32 (1.14)
  post-test (9 months): number analyzed (Participants) | 50 | 46
  post-test (9 months) | 8.8 (1.37) | 9.17 (1.06)
  6 month follow-up (6-month post intervention completion) | 9.16 (1.33) | 9.21 (1.25)

14. Secondary Outcome: Self-Esteem
Description: Self-esteem was measured using the Rosenberg Self-Esteem Scale (RSES) (Rosenberg, 1965). The scale is a common measure of self-esteem (Sinclair et al., 2010) and has been used across different cultural contexts with high internal consistency, including in Ghana (α = 0.83-0.85) (Ahulu et al., 2020; Glozah, 2014). The scale comprises 10 statements about general feelings of self-worth or self-acceptance rated on a 4-point Likert scale response option (strongly agree to strongly disagree, with 4 = strongly agree, 3 = agree, 2 = disagree, 1 = strongly disagree). The items were scored on a theoretical range of 10-40 and summed, with higher scores representing higher self-esteem.
Time Frame: baseline, post-test (9 months), 6 month follow-up (6-month post intervention completion)
Population: Adolescent girls. One participant was lost to follow-up at 9 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 50
score on a scale
  6 month follow-up | 34.02 (3.58) | 33.48 (4.34)
  post-test (9 months): number analyzed (Participants) | 46 | 50
  post-test (9 months) | 33.15 (2.80) | 32.78 (5.51)
  Baseline | 29.96 (4.55) | 31.3 (4.10)

15. Secondary Outcome: Emotional Self-efficacy
Description: Emotional self-efficacy was assessed using the Emotional self-efficacy scale (ESE; Valois & Zulig, 2013), an 8-item scale to measure an individual's perceived ability to manage emotions effectively. This scale has been widely used to evaluate emotional self-regulation across different contexts. Participants responded to each item on a 5-point Likert scale ranging from 1 (not at all well) to 5 (very well) (theoretical range 8-40). Sample items included, "How well do you succeed in cheering yourself up when an unpleasant event has happened?" and "How well do you succeed in becoming calm again when you are very scared?" Scores were summed, with higher scores reflecting greater emotional self-efficacy
Time Frame: baseline, post-test (9 months), 6-month follow-up (15 months)
Population: At 9 months follow-up, one person was lost during interviews in the treatment arm. However, this participants was interviewed at 15 months follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Bolstered Care | Anzansi Family Program
Number analyzed (Participants) | 50 | 47
score on a scale
  baseline | 31.44 (4.99) | 30.53 (7.10)
  post-test (9 months): number analyzed (Participants) | 50 | 46
  post-test (9 months) | 29.44 (6.33) | 33.91 (4.97)
  6-month follow-up (15 months) | 32.28 (6.95) | 33.94 (4.96)

16. Secondary Outcome: Social Self-efficacy
Description: Social self-efficacy was measured using the Social self-efficacy scale (Zullig, Teoli, Valois, 2011), a 8-item scale to evaluate an individual's confidence in handling social situations and interactions. Participants rated their responses on a 5-point Likert scale, ranging from 1 (not at all well) to 5 (very well). Sample items included "How well can you express your opinions when other classmates disagree with you?" and "How well can you become friends with other children?" The items were summed, with higher scores indicating greater social self-efficacy (theoretical range 8-40).
Time Frame: baseline, post-test (9 months), 6-month follow-up (15 months)
Population: One participant was lost to follow-up at 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Bolstered Care | Anzansi Family Program
Number analyzed (Participants) | 50 | 47
score on a scale
  baseline | 32.32 (4.44) | 32.51 (4.86)
  post-test (9 months): number analyzed (Participants) | 50 | 46
  post-test (9 months) | 30.18 (6.38) | 35.54 (4.12)
  6-month follow-up (15 months | 34.32 (5.68) | 36.62 (3.75)

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Control: Bolstered Care | Anzansi Family Program
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/94
Other Adverse Events (participants affected / at risk) | 0/100 | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT04231669/Prot_SAP_000.pdf